CLINICAL TRIAL: NCT05143034
Title: Evaluation of Skin Efficacy of TCI66207
Brief Title: the Evaluation of the Efficacy of TCI66207 on the Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSMH No.18-148-A
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCI66207 Essence (Experimental): Essence
  Interventions: Dietary Supplement: TCI66207 Essence
- Placebo Essence (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Essence

INTERVENTIONS:
Dietary Supplement: TCI66207 Essence — Use it twice a day after washing your face in the morning and evening for a total of 4 weeks.
  Arms: TCI66207 Essence
Dietary Supplement: Placebo Essence — Use it twice a day after washing your face in the morning and evening for a total of 4 weeks.
  Arms: Placebo Essence

SUMMARY:
The purpose of this study is to explore the evaluation of the efficacy of TCI66207 deep-sea live-face bacteria on the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged above 20 years old
2. Subject has dull skin.

Exclusion Criteria:

1. .Subject with diseases of the skin, heart, liver, kidney, endocrine and other organs and patients with mental illness (according to medical history).
2. Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
3. Female who is pregnant or nursing or planning to become pregnant during the course of the study.
4. Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
5. Subjects who have large spots (area >3 square centimeter) or abnormal acne.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of skin moisture | Subjects will be tested in the 4th week.
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin elasticity | Subjects will be tested in the 4th week.
  Cutometer® dual MPA 580 was utilized to measure skin elasticity (parameter R2). Units: μm penetration depth into the probe opening, expressed as curvesCorneometer® units 0-120
The change of skin wrinkles | Subjects will be tested in the 4th week.
  VISIA Complexion Analysis System was utilized to measure wrinkles. Units: arbitrary units
The change of skin collagen density | Subjects will be tested in the 4th week.
  DermaLab® USB - 20 MHz High Freq. Ultrasound probe was utilized to scan and analyze skin collagen density. Units: Intensity score
The change of skin texture | Subjects will be tested in the 4th week.
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Subjects will be tested in the 4th week.
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Research & Design Center, TCI CO., Ltd, Taipei, Neipu Township, Taiwan